CLINICAL TRIAL: NCT07187089
Title: An Open-Label, Single-Arm Study to Assess Growth and Bone Mineral Density in Children ≥6 to <12 Years of Age With Severe Atopic Dermatitis Treated With Dupilumab
Brief Title: Study of Growth and Bone Mineral Density in Children With Atopic Dermatitis (AD) Treated With Dupilumab
Acronym: BUILD-PEDS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-2372
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Severe Atopic Dermatitis (AD)
Keywords: Uncontrolled AD; Bone Mineral Accrual (BMA); Bone growth; Shorter stature; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dupilumab (Experimental)
  Interventions: Drug: dupilumab

INTERVENTIONS:
Drug: dupilumab — Administered per the protocol
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
This study is researching an approved drug called dupilumab (called "study drug"). Dupilumab is approved in the United States for the treatment of adult and pediatric patients aged 6 months and older with moderate-to-severe atopic dermatitis (also commonly known as eczema).

The aim of the study is to see if dupilumab treatment of children with severe atopic dermatitis, which cannot be adequately controlled with topical atopic dermatitis medication, improves growth and bone strength.

The study is looking at other research questions, including:

• What side effects may happen from taking dupilumab

ELIGIBILITY:
Key Inclusion Criteria:

1. Children with body weight ≥15 kg and <60 kg at screening visit 1
2. Diagnosis of AD according to American Academy of Dermatology consensus criteria at time of screening visit
3. Investigator Global Assessment (IGA) score = 4 at screening and baseline visits
4. ≥15% Body Surface Area (BSA) of AD involvement at the screening and baseline visits
5. Worst Itch Scale score ≥4 at screening visit (for prior 24 hours) and baseline visit (weekly average over prior 7 days)
6. Shorter stature defined for the study as ≤30th height-for-age percentile at screening, as defined in the protocol
7. AD not adequately controlled with topical corticosteroid prescription therapies or when those therapies are not advisable, as defined in the protocol

Key Exclusion Criteria:

1. Females who have passed menarche at screening
2. Concomitant skin diseases that may confound AD assessments in the opinion of the investigator
3. Has a known medical issue which may contribute to shorter stature (eg, growth hormone deficiency, Celiac disease)
4. Active helminthic infections; suspected or high risk of helminthic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before baseline
5. Has a known allergy or hypersensitivity to components of the study intervention
6. Prior use of dupilumab or other biologic treatment for AD, as defined in the protocol
7. Other advanced systemic treatment for AD within 4 weeks or non-steroidal topical treatments within 2 weeks before the baseline visit

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria Apply

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-11-11 (Estimated); Primary Completion 2027-12-23 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of ≥5 percentile in height-for-age percentile on the Centers for Disease Control and Prevention (CDC) growth chart | Baseline to Week 52
  The Centers for Disease Control and Prevention (CDC) growth charts use percentile scales as a measurement system. The percentile scale is a ranking system that compares a child's growth measurements (e.g., height, weight, Body Mass Index [BMI]) to a reference population of the same age and sex.

SECONDARY OUTCOMES:
Change from baseline in Lumbar Spine (LS) Bone Mineral Density (BMD) adjusted Z-score measured by Dual-Energy X-Ray Absorptiometry (DEXA) | Baseline to Week 52
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through Week 54
Occurrence of Serious Adverse Events (SAEs) | Through Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/